CLINICAL TRIAL: NCT06713421
Title: The Effects of Premedication With Pronase and Postural Exercise on Mucosal Cleanliness During Painless Esophagogastroduodenoscopy: A Prospective, Multicenter, Randomized Controlled Study Based on Artificial Intelligence Assessment
Brief Title: Effect of Premedication With Pronase on Mucosal Cleanliness During EGD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Fujian Provincial Hospital (Other); Huashan Hospital (Other); The Second Affiliated Hospital of Harbin Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Red Cross Hospital, Hangzhou, China (Other); The Affiliated Hospital of Inner Mongolia Medical University (Other); Yuebei People's Hospital (Other); Longgang District People's Hospital of Shenzhen (Other); Huadu District People's Hospital of Guangzhou (Other); Liaocheng People's Hospital (Other); Qilu Hospital of Shandong University (Other); The Second Affiliated Hospital of Shandong First Medical University (Other); Anqing Municipal Hospital (Other); Jiujiang No.1 People's Hospital (Other); Kunshan Hospital of Traditional Chinese Medicine (Unknown); Nanjing Gaochun People's Hospital (Other); Taizhou First People's Hospital (Other); Hengshui People's Hospital (Other); Affiliated Hospital of Hebei University (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Taihe Hospital (Other); ZhuZhou Central Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); Subei People's Hospital of Jiangsu Province (Other); The Affiliated Hospital Of Southwest Medical University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Loudi Central Hospital (Other); Beijing Tiantan Hospital (Other); Peking Union Medical College Hospital (Other); The First People's Hospital of Lin'an District, Hangzhou (Unknown); Zhejiang Provincial People's Hospital (Other); Jining Medical University (Other); Ningbo Medical Center Lihuili Hospital (Other Government); Zhoushan Hospital, Zhejiang (Unknown); General Hospital of Ningxia Medical University (Other); Yunnan Cancer Hospital (Other); Xinghua City People's Hospital (Unknown); Beijing Friendship Hospital, Captial Medical University (Unknown); Beijing Chao-Yang Hospital, Captial Medical University (Unknown); The People's Hospital of JiangMen (Unknown); The First People's Hospital of TianMen in Hubei Province (Unknown); THE FIRST AFFILIATED HOSPITAL OF SHIHEZI UNIVERSITY (Unknown)
Responsible Party: Principal Investigator, Luowei Wang, MD, Clinical Professor, Changhai Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: EPPMC
Record Dates: First submitted 2024-11-09; First posted 2024-12-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: EGD; Pronase; Postural exercise; Mucosal cleanliness
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — dimethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- A1:Dimeticone+Pronase+Postural Exercise group (Experimental): Approximately 15-20 minutes before EGD, patients orally receive 50mL of warm water containing 5g dimethicone powder and 20,000 IU pronase granules combined with 1 g NaHCO3. Then the patients are asked to take a 3-minute postural exercise.
  Interventions: Drug: Dimethicone+Pronase; Behavioral: with Postural Exercise
- A2:Dimeticone+Pronase group (Experimental): Approximately 15-20 minutes before EGD, patients orally receive 50mL of warm water containing 5g dimethicone powder and 20,000 IU pronase granules combined with 1 g NaHCO3. Then the patients sit quietly awaiting examination.
  Interventions: Drug: Dimethicone+Pronase; Behavioral: without Postural Exercise.
- B1:Dimeticone+Postural Exercise group (Active Comparator): Approximately 15-20 minutes before EGD, patients orally receive 50mL of warm water containing 5g dimethicone powder. Then the patients are asked to take a 3-minute postural exercise.
  Interventions: Drug: Dimethicone; Behavioral: with Postural Exercise
- B2:Dimeticone group (Active Comparator): Approximately 15-20 minutes before EGD, patients orally receive 50mL of warm water containing 5g dimethicone powder. Then the patients sit quietly awaiting examination.
  Interventions: Drug: Dimethicone; Behavioral: without Postural Exercise.

INTERVENTIONS:
Drug: Dimethicone+Pronase — Approximately 15-20 minutes before EGD, patients orally receive 50mL of warm water containing 5g dimethicone powder and 20,000 IU pronase granules combined with 1 g NaHCO3.
  Arms: A1:Dimeticone+Pronase+Postural Exercise group; A2:Dimeticone+Pronase group
Drug: Dimethicone — Approximately 15-20 minutes before EGD, patients orally receive 50mL of warm water containing 5g dimethicone powder.
  Arms: B1:Dimeticone+Postural Exercise group; B2:Dimeticone group
Behavioral: with Postural Exercise — After the premedication is administered orally approximately 15-20 minutes before EGD, patients are asked to take a 3-minute postural exercise.
  Arms: A1:Dimeticone+Pronase+Postural Exercise group; B1:Dimeticone+Postural Exercise group
Behavioral: without Postural Exercise. — After the premedication is administered orally approximately 15-20 minutes before EGD, patients sit quietly awaiting examination.
  Arms: A2:Dimeticone+Pronase group; B2:Dimeticone group

SUMMARY:
Gastric cancer and esophageal cancer are common malignant tumors that threaten people's life and health. Esophagogastroduodenoscopy (EGD) is an important tool for screening upper gastrointestinal tumors, especially early tumors, and an effective method for detecting other upper gastrointestinal lesions, including ulcers and polyps. However, during EGD examination, mucus and foam can reduce the cleanliness of the mucosa and limit the operator's visual field, resulting in missed lesions and misdiagnosis. Previous studies have shown that preoperative medication with pronase and dimeticone is correlated with the improvement of upper gastrointestinal mucosal cleanliness. However, the number of samples in such studies is limited, and the artificial judgment is not objective enough to evaluate the cleanliness of upper digestive tract mucosa. And, whether a postural exercise is necessary for premedication with pronase or dimeticone remains unclear. Our team design this experiment to examine the efficacy of using premedication of dimeticone/pronase with a postural exercise on visualization of the mucosa before painless EGD. The investigators aim to provide new evidence to optimize the use of premedication with EGD.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years and ≤70 years;
2. Voluntarily participate in the trial and sign the informed consent.

Exclusion Criteria:

1. active gastrointestinal bleeding;
2. esophageal stricture, complete pyloric obstruction and gastroparesis caused by various reasons;
3. diagnosed malignant tumors of the upper digestive tract;
4. a history of upper gastrointestinal surgery;
5. severe heart, liver and kidney diseases, and the doctor judges that it is not suitable for painless gastroscopy;
6. serious mental illness;
7. pregnancy or breastfeeding;
8. an allergy to pronase or dimeticone;
9. current participation in other clinical trials and in the follow-up or drug washout period;
10. patients considered by the investigator to be unsuitable for this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Mucosal Cleanliness Scores | Through study completion, an average of 1 year
  The upper digestive tract is divided into 9 anatomical parts, including esophagus, squamocolumnar junction, middle-upper gastric body, lower gastric body, gastric antrum, duodenal bulb, duodenal descending, gastric angulus and gastric fundus.
  The mucosal cleanliness score of each segment is classified as 0-3. Score0: any solid food, blood or blood clots, or other content that could not be suctioned or washed, or an obstruction that prevented adequate visualization of the majority of an anatomical area.
  Score 1: mucus, bubbles, liquid content, and blood that required suctioning AND/OR washing.
  Score 2: nonadherent liquid content or blood that required ONLY suctioning but NOT washing.
  Score 3: entire mucosa well seen without the need for suctioning or washing. The sum of the mucosal cleanliness scores for the above mentioned 9 locations ranges from 0 to 27.

SECONDARY OUTCOMES:
Procedure Time | Through study completion, an average of 1 year
  The procedure time of EGD is defined as the time taken from the entry of EGD into the esophagus to the withdrawal of the EGD.
The Detection Rate of Diminutive Lesions | Through study completion, an average of 1 year
  The detection rate of diminutive lesions means the proportion of patients with diminutive lesions <5 mm.
Safety of antifoam/mucus agents | Through study completion, an average of 1 year
  Any adverse event including gag reflex and hypoxemia during EGD examination need to be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Luowei Wang, MD, Principal Investigator — Changhai hosipital, Shanghai
Locations (1):
- Changhai hosipital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No